CLINICAL TRIAL: NCT00336089
Title: The Effects of Cross Training on Fatigue and Pain Levels in Breast Cancer Survivors
Brief Title: Exercise Program or Health Education Program in Reducing Fatigue and Pain in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clayton State University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: CDR0000466676; CSU-GCC-161
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer; Cancer Survivor; Fatigue; Pain
Keywords: fatigue; pain; cancer survivor; breast cancer in situ; inflammatory breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Pain; Breast Carcinoma In Situ; Inflammatory Breast Neoplasms | interventions — Early Intervention, Educational; Therapeutics; Analgesia

INTERVENTIONS:
Behavioral: exercise intervention
Other: educational intervention
Procedure: complementary or alternative medicine procedure
Procedure: fatigue assessment and management
Procedure: management of therapy complications
Procedure: pain therapy
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: An exercise program or health education program may help relieve fatigue and pain and improve the quality of life in women who are breast cancer survivors. It is not yet known whether an exercise program is more effective than a health education program or no program in reducing fatigue and pain in women who are breast cancer survivors.

PURPOSE: This randomized clinical trial is studying an exercise program to see how well it works in reducing fatigue and pain compared to a health education program or no program in women who are breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether a moderate-intensity exercise program comprising cardiorespiratory and resistance training of the legs, back, abdominal, trunk, and arm musculature vs a control group attenuates fatigue and pain in breast cancer survivors.
* Determine whether this exercise program will significantly improve the quality of life of these patients.
* Determine whether this exercise program can significantly reduce the number of days of absenteeism from work in these patients.
* Determine whether this exercise program can significantly attenuate mood disturbances in these patients.

OUTLINE: This is a randomized, controlled, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (exercise program): Patients participate in an exercise program comprising cardiorespiratory (walking on a treadmill) and resistance training for 1 hour, 3 times weekly for 12 weeks.
* Arm II (control): Patients undergo no intervention. In both arms, patients complete questionnaires regarding general health, mood, work attendance, and physical activity before the start of study treatment and then every 3 weeks for 12 weeks. Patients also complete a 7-day physical activity diary and sleep diary every 3 weeks.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Breast cancer survivor
* Received adjuvant chemotherapy or radiotherapy for breast cancer only

  * Must have completed treatment 2-6 months ago
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Hemoglobin ≥ 11 g/dL
* Able to read English
* No high-risk for cardiovascular problems during exercise, including any of the following:

  * Unstable heart disease
  * Unstable angina
  * Chronic respiratory disease
  * Dizziness
  * Uncontrolled hypertension
* No severe respiratory disease requiring oxygen therapy
* No history of anorexia (body mass index [BMI] < 18.5) or severe obesity (BMI > 35)
* No history of multiple cancers
* No shortness of breath or hypotension
* No sudden swelling of the ankles, hands or face
* No palpitations or arrhythmias
* No persistent and intolerable pain
* No major acute illness (e.g., fever or respiratory infection)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Poudevigne, PhD, Study Chair — Clayton State University
Locations (2):
- United States (2):
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Clayton State University, Morrow, Georgia